CLINICAL TRIAL: NCT05858346
Title: A Randomized Clinical Trial Comparing Transdiagnostic Behavior Therapy to Disorder-Specific Psychotherapy in the Recovery of Veterans With Social Anxiety Disorder and Comorbid PTSD Symptomatology
Brief Title: Comparing TBT to Disorder-Specific Psychotherapy in Veterans With Social Anxiety Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D4516-R
Record Dates: First submitted 2023-04-25; First posted 2023-05-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transdiagnostic Behavior Therapy (Experimental): TBT was developed to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and [positive] emotional/behavioral activation). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders.
  Interventions: Behavioral: Transdiagnostic Behavior Therapy
- Cognitive Behavioral Therapy for Social Anxiety Disorder (Active Comparator): To provide an evidence-based comparison for the TBT condition, the research-supported psychological treatment of CBT for SAD will be used. CBT for SAD demonstrates efficacy in improving SAD symptoms and quality of life for patients with SAD, with durable improvements evidenced at follow-up assessments. CBT for SAD was used as a comparison to TBT in previous preliminary research. CBT for SAD involves several primary components, including: 1) psychoeducation, 2) training in cognitive restructuring, 3) exposures, 4) advanced cognitive restructuring, and 5) termination.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Social Anxiety Disorder

INTERVENTIONS:
Behavioral: Transdiagnostic Behavior Therapy — TBT was developed to address transdiagnostic avoidance via the use of four different types of exposure techniques (situational/in-vivo, physical/interoceptive, thought/imaginal, and [positive] emotional/behavioral activation). From the transdiagnostic avoidance perspective, the four exposure practices are matched to the type(s) of avoidance experienced by patients based upon their cluster of symptoms/disorders.
  Arms: Transdiagnostic Behavior Therapy
Behavioral: Cognitive Behavioral Therapy for Social Anxiety Disorder — To provide an evidence-based comparison for the TBT condition, the research-supported psychological treatment of CBT for SAD will be used. CBT for SAD demonstrates efficacy in improving SAD symptoms and quality of life for patients with SAD, with durable improvements evidenced at follow-up assessments. CBT for SAD was used as a comparison to TBT in previous preliminary research. CBT for SAD involves several primary components, including: 1) psychoeducation, 2) training in cognitive restructuring, 3) exposures, 4) advanced cognitive restructuring, and 5) termination.
  Arms: Cognitive Behavioral Therapy for Social Anxiety Disorder

SUMMARY:
Cognitive behavioral therapy (CBT) is a brief, efficient, and effective treatment for individuals with depressive/anxiety disorders. However, CBT is largely underutilized within the Department of Veterans Affairs due to the cost and burden of trainings necessary to deliver all of the related disorder-specific treatments (DSTs). Transdiagnostic Behavior Therapy (TBT), in contrast, is specifically designed to address numerous distinct disorders within a single protocol in Veterans with depressive/anxiety disorders. The proposed research seeks to evaluate the efficacy of TBT by assessing psychiatric symptomatology and related impairment outcomes in Veterans with social anxiety disorder and comorbid posttraumatic stress via a randomized controlled trial of TBT and an existing DST. Assessments will be completed at pre-, mid-, and post-treatment, and at 6-month follow-up. Process variables also will be investigated.

DETAILED DESCRIPTION:
Objective The objective of the present study is to examine efficacy of TBT in improving quality of life, psychological well-being, and social reintegration of Veterans with SAD and comorbid PTSD symptomatology compared to a DST for SAD using an RCT design. Patient satisfaction and predictors of feasibility (attendance and discontinuation) also will be assessed.

Recruitment Strategy Veterans will be recruited through the Primary Care Mental Health Integration, General Outpatient Mental Health, and Mental Health Specialty Clinic (e.g., PTSD Clinical Team) programs within the Charleston VAHCS and associated CBOCs. Within the targeted clinics, all Veterans reporting symptoms of social anxiety meet with a mental health staff member to complete a clinical interview and self-report measures. If Veterans endorse symptoms consistent with SAD and PTSD symptomatology, interest in participating in research will be assessed and, if agreeable, the Veteran will be referred to project staff.

Intake Procedures A study-specific intake appointment will be completed with the project staff to complete consent documentation as well as assess inclusion and exclusion criteria, including a semi-structured clinical interview and self-report questionnaires. Screening and consent will take place at the participant's residence via telehealth by research staff or in person at the VAHCS, based upon the preference of the participant.

Treatment Procedures Participants who meet inclusion and exclusion criteria will be randomized into a study condition and assigned to a project therapist. Eligible VAHCS patients will be randomized into one of two treatment conditions: TBT or DST (CBT for SAD). Both treatment conditions will include 12 weekly 60-minute individual psychotherapy sessions. The general format of sessions will involve: 1) brief check-in; 2) review of materials from previous sessions; 3) review of homework assignments; 4) overview of new materials and in-session exercises; and 5) assignment of homework for next session. Attendance and homework completion will be recorded.

Randomization Procedures Participants will be randomly assigned (1:1) to one of the two study arms using a permuted block randomization procedure. After determining eligibility and completing consent and baseline assessment materials, enrolled participants will be assigned to treatment conditions using a computer-generated randomization scheme and communicated to the assigned study therapist. Once randomized, participants will be included in the intent-to-treat analysis. Randomization will occur at the participant level.

Treatment Training and Fidelity All therapy will be led by one of the project therapists in a rotating fashion. Training workshops will be provided for the two treatment protocols. Established trainers and experts will be recruited to provide each of the trainings. Trainings will be supported by weekly supervision on the two protocols led by the matching trainer throughout the duration of the treatment phase, with additional supervision sessions provided as needed.

Consistent with other well-designed treatment outcome studies, all treatment sessions will be audio recorded with 20% of sessions randomly selected for review for treatment integrity and fidelity. These integrity and fidelity reviews will focus on evaluating the match between the treatment manuals and the material covered in session. To evaluate adherence, treatment-specific rating forms will be used to determine if the therapist appropriately covered the content of each session. Experts will be recruited to rate the recordings independently, with feedback provided to the therapists throughout the duration of the study to maintain treatment delivery with high fidelity.

Assessment of Quality of Life, Psychological Well-Being, Social Reintegration, Psychiatric Symptomatology, and Treatment Satisfaction Follow-up assessments will be conducted for all participants during VA visits or via home based telehealth by trained interviewers blind to treatment conditions. The battery of self-report questionnaires and a diagnostic interview will be completed pre-, mid-, and post-treatment and at the 6-month follow-up to track participant progress through the treatment and maintenance phases.

To reduce the likelihood of missing data, primary assessments will be scheduled separately from treatment sessions. The biweekly measures will include disorder-specific measures that will be administered at the beginning of therapy sessions and used to inform the clinical delivery of the psychotherapies (measurement-based care) and assist in the intent-to-treatment analyses and analysis of trajectories.

All assessments will be completed by the Project Research Recruiter and Assessor. Additional training will be required prior to administration of the diagnostic interview. The assessor will be blinded to treatment condition and supervised by the PI. Assessments will be recorded to investigate inter-rater reliability of diagnoses, with 20% of recordings being re-assessed by a trained assessor after the participant has completed all study procedures, with feedback provided to the assessor throughout the study to maintain high reliability.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be Veterans and registered at Ralph H. Johnson Veterans Affairs Health Care System
* Participants must be clearly competent to provide informed consent for research participation
* Participants must meet DSM-5 criteria for social anxiety disorder
* Participants must have clinically significant symptoms of comorbid posttraumatic stress

Exclusion Criteria:

* recent history (< 2 months) of psychiatric hospitalization or a suicide attempt as documented in their medical record,
* acute, severe illness or medical condition that likely will interfere with study procedures as documented in their medical record
* recent start of new psychiatric medication(s) (< 4 weeks),
* primary diagnosis of a condition associated with psychotic symptoms, personality disorder, substance use disorder, or bipolar disorder.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
MASA functional impairment | change from baseline to week 6 to week 12 to 6-month followup
  The MASA is a 38-item self-report measure that was designed to assess trait symptom dimensions consistent with the hybrid model of social anxiety. The MASA contains six subscales that assess behavioral avoidance, physiological arousal and avoidance, thought avoidance, anhedonia, functional impairment, and coping with substances. The six subscales have shown to differentiate symptoms across anxiety disorders and depression and their comorbidities and to be sensitive to improvements evidenced in therapy.
PTSD Checklist for DSM-5 (PCL-5) | change from baseline to week 6 to week 12 to 6-month followup
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses DSM-5 criteria PTSD symptoms. Items are scored on a 5-point scale, range from 0 (not at all) to 4 (extremely). The total scale score ranges from 0 to 80 with higher scores associated with more severe symptomatology. Previous versions of the PCL have been shown to have excellent internal consistency and excellent test-retest reliability in Veterans. In addition, the PCL-5 has been incorporated into standard assessment for PTSD at the VA. The PCL5 will be used to assess symptoms of PTSD.
Illness Intrusiveness Rating Scale (IIRS) | change from baseline to week 6 to week 12 to 6-month followup
  The IIRS is a 13-item questionnaire that assesses the extent to which a disease interferes with important domains of life, including health, diet, work, and several others. The IIRS has been shown to have strong psychometric properties in the previous literature in participants with physical and emotional health concerns, and has been used in previous TBT studies.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Gros, PhD MA BS, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon consultation with the local VA R&D and MUSC IRB committees after publication of primary research questions, the de-identified database will be made available to the public via the publishing journal's website (where applicable) as well as on (yet to be determined/selected) research community websites designed for the sharing of scientific findings and data.
Supporting Information: Study Protocol
Time Frame: starting 6 months after publication of the primary outcome papers